CLINICAL TRIAL: NCT04248543
Title: Quantitative MR Imaging Methods for Functional Assessment Following Stereotactic Body Radiation Therapy for Spinal Metastases
Brief Title: Quantitative MRI for Functional Assessment Following SBRT for Spinal Metastases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: Pro00103960
Record Dates: First submitted 2020-01-23; First posted 2020-01-30 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Spinal Metastases
Keywords: Vertebral compression fracture; Radiation induced myelopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- quantitative MRI at 4 weeks (Experimental)
  Interventions: Device: qMRI with Gadoteridol contrast agent

INTERVENTIONS:
Device: qMRI with Gadoteridol contrast agent — quantitative MR: MRI uses a magnet and radio waves to make medical images of the body. Gadoteridol is used as a contrast agent. Quantitative MRI involves the use of software to analyze the acquired images.
  Other Names: quantitative MRI

SUMMARY:
The purpose of this study is to determine if quantitative magnetic resonance imaging (qMRI) can objectively measure changes in the tumor/vertebral body and adjacent spinal cord following stereotactic body radiation therapy (SBRT) for painful metastatic spine disease.

DETAILED DESCRIPTION:
Metastatic spine disease (MSD) can result in considerable morbidity from pain, spinal cord compromise and neurologic disability. Recent developments in image-guidance and immobilization have enabled more accurate target localization, which allows methods of precise high-dose radiation delivery such as stereotactic body radiation therapy (SBRT). SBRT carries potential risks of radiation induced myelopathy (RIM) and vertebral compression fracture (VCF). Magnetic resonance imaging (MRI) is a sensitive imaging modality that may be able to detect radiation-induced damage in the vertebral body or spinal cord following SBRT. Quantitative MR-based imaging methods may also help to quantify treatment response and help predict subsequent outcomes such as tumor control and VCF risk.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of metastatic cancer with a vertebral body metastasis or contiguous vertebral body metastases for which SBRT is appropriate
* Age ≥ 18 years of age
* KPS ≥ 70
* Life expectancy of at least 3 months
* No contraindication to undergoing MR imaging
* Women of childbearing age must have a negative urine or serum pregnancy test to meet eligibility per Duke Policy
* Pre-treatment pain score of at least 1/10 based on the numeric pain rating scale (NPRS)
* Disease located from C1 to S5
* Subjects with prior radiation to the involved vertebral body are allowed.

Exclusion Criteria:

* Subjects unable to undergo MRI (includes non-MRI compatible material or devices and severe claustrophobia)
* Subjects with prior procedural intervention to the involved vertebral body that would result in artifact (kyphoplasty, screw and/or rod placement); minimally invasive surgery without instrumentation of the involved vertebral body and instrumentation immediately above or below the index lesion is allowed.
* Subjects with spinal cord compression; minimally invasive "separation" surgery to first resect the epidural component is allowed
* Pregnant or breast-feeding women
* Allergy to standard IV contrast agents used in MRI
* Subjects with eGFR <30 30 mL/min2 or on dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-12-22 (Actual); Primary Completion 2025-07-02 (Actual); Study Completion 2025-07-02 (Actual)

PRIMARY OUTCOMES:
Relative Change in Sequence specific parameters for Diffusion tensor imaging (DTI) | baseline, 4 wks
Relative Change in Sequence specific parameters for Diffusion weighted imaging (DWI) | baseline, 4 wks
Relative Change in Sequence specific parameters for Dynamic contrast enhanced (DCE) MRI | baseline, 4 wks

SECONDARY OUTCOMES:
Change in numeric pain score as measured by the Numeric Pain Rating Scale | baseline, 4 wks
  Measured from 0-10 with 0 being no pain and 10 being severe pain
Change in numeric pain score as measured by the Brief Pain Inventory | baseline, 4 wks
  Measured from 0-10 with 0 being no pain and 10 being worst imaginable pain
Change in numeric pain score as measured by the EQ5D Pain Questionnaire | baseline, 4 wks
  Measured from 0-10 with 0 being no pain and 10 being worst imaginable pain
Change in opioid use | baseline, 4 wks
Change in quality of life as measured by the Pat Sf36 V2 assessment | baseline, 4 wks
  Pat SF36 V2 is a quality of life survey about physical activity, general health and daily functions measured from excellent/much better/yes, limited a lot/all of the time/not at all, through poor/much worse/no,not limited at all/none of the time/extremely with additional not answered option
Change in quality of life as measured by the PROMIS assessment | baseline, 4 wks
  PROMIS categories include physical function, anxiety, depression, fatigue, sleep and pain ranging from never/not at all through always/very much.
Change in quality of life as measured by the SOSG+ assessment | baseline, 4 wks
  Questionnaire about physical function, neurological function and pain ranging from never/not at all through always/very much

CONTACTS AND LOCATIONS:
Overall Officials: Trey Mullikin, MD, Principal Investigator — Duke University
Locations (1):
- Duke Cancer Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No